CLINICAL TRIAL: NCT00509496
Title: Phase II Study of Metastatic Melanoma Using Lymphodepleting Conditioning Followed by Infusion of Anti-gp100:154-162 TCR-Gene Engineered Lymphocytes
Brief Title: Phase II Study of Metastatic Melanoma With Lymphodepleting Conditioning and Anti-gp100:154-162 TCR Gene Engineered Lymphocytes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070174; 07-C-0174
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2012-12

CONDITIONS: Skin Cancer; Melanoma
Keywords: Refractory; Gene Therapy; HLA-A2 Positive; Stage IV Melanoma; Melanoma; Skin Cancer; Malignant Melanoma
MeSH Terms: conditions — Skin Neoplasms; Melanoma | interventions — fludarabine phosphate; Cyclophosphamide; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anti-gp100:154-162 TCR PBL + HD IL-2 (Experimental): 1. fludarabine phosphate-25 mg/m^2/day intravenous piggy back over 30 minutes for 5 days
  2. cyclophosphamide-60 mg/kg/day x 2 days intravenous
  3. Anti-gp100:154-162 TCR-engineered peripheral blood lymphocyte (PBL) cell preparation - minimum of approximately 5 X 10^8 cells and up to 3 x10^11 anti-gp100:154-162 TCR engineered TIL or PBL. The cells are infused intravenously over 20-30 minutes.
  4. aldesleukin-720,000 IU/kg intravenously over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses)
  Interventions: Drug: fludarabine phosphate; Drug: cyclophosphamide; Biological: aldesleukin; Biological: autologous anti-gp 100:154-162 T-cell receptor gene-engineered peripheral blood lymphocytes
- anti-gp100:154-162 TCR TIL + HD IL-2 (Experimental): 1. fludarabine phosphate-25 mg/m^2/day intravenous piggy back over 30 minutes for 5 days
  2. cyclophosphamide-60 mg/kg/day x 2 days intravenous
  3. Anti-gp100:154-162 TCR-engineered tumor infiltrating lymphocytes (TIL) cell preparation- minimum of approximately 5 X 10^8 cells and up to 3 x10^11 anti-gp100:154-162 TCR engineered TIL or PBL. The cells are infused intravenously over 20-30 minutes
  4. aldesleukin-720,000 IU/kg intravenously over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses)
  Interventions: Drug: fludarabine phosphate; Drug: cyclophosphamide; Biological: aldesleukin; Biological: autologous anti-gp 100:154-162 T-cell receptor gene-engineered tumor infiltrating lymphocytes

INTERVENTIONS:
Drug: fludarabine phosphate — 25 mg/m^2/day intravenous piggy back over 30 minutes for 5 days.
  Other Names: Fludara
Drug: cyclophosphamide — 60 mg/kg/day x 2 days intravenous
  Other Names: Cytoxan
Biological: aldesleukin — 720,000 IU/kg intravenously over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses).
  Other Names: IL-2
Biological: autologous anti-gp 100:154-162 T-cell receptor gene-engineered tumor infiltrating lymphocytes — Patients will receive a minimum of approximately 5 X 10^8 cells and up to 3 x10^11 anti-gp100:154-162 TCR engineered TIL .
  The cells are infused intravenously over 20-30 minutes.
  Arms: anti-gp100:154-162 TCR TIL + HD IL-2
Biological: autologous anti-gp 100:154-162 T-cell receptor gene-engineered peripheral blood lymphocytes — Patients will receive a minimum of approximately 5 X 10^8 cells and up to 3 x10^11 anti-gp100:154-162 TCR engineered PBL.
  The cells are infused intravenously over 20-30 minutes.
  Arms: anti-gp100:154-162 TCR PBL + HD IL-2

SUMMARY:
Background:

* Human peripheral blood lymphocytes have been engineered to express a T-cell receptor (TCR) that recognizes a blood type, human leukocyte antigen (HLA-A*0201) derived from the gp100 protein. A retroviral vector was constructed that can deliver the TCR to cells.
* This gene-engineered cell is over 10 times more reactive with melanoma cells than is the melanoma antigen recognized by T-cells (MART-1) TCR that resulted in tumor shrinkage for two patients with metastatic melanoma.

Objectives:

* To determine whether an anti-melanoma protein receptor can be put in cells removed from patients' tumors or blood and then reinfused, with the purpose of shrinking tumors.
* To evaluate safety and effectiveness of the treatment.

Eligibility:

* Patients 18 years of age or older with metastatic cancer melanoma (cancer that has spread beyond the original site).
* Patient's leukocyte antigen type is HLA-A*0201.

Design:

-Patients undergo the following procedures:

* Leukapheresis (on two occasions). This is a method of collecting large numbers of white blood cells. The cells obtained in the first leukapheresis procedure are grown in the laboratory, and the anti-gp100 protein is inserted into the cells using an inactivated (harmless) virus in a process called retroviral transduction. Cells collected in the second leukapheresis procedure are used to evaluate the effectiveness of the study treatment.
* Chemotherapy. Patients are given chemotherapy through a vein (intravenously, IV) over 1 hour for 2 days to suppress the immune system so that the patient's immune cells do not interfere with the treatment.
* Treatment with anti-gp100. Patients receive an IV infusion of the treated cells containing anti-gp100 protein, followed by infusions of a drug called IL-2 (aldesleukin), which helps boost the effectiveness of the treated white cells.
* Patients are given support medications to prevent complications such as infections.
* Patients may undergo a tumor biopsy (removal of a small piece of tumor tissue).
* Patients are evaluated with laboratory tests and imaging tests, such as CT scans, 4 to 6 weeks after treatment and then once a month for 3 to 4 months to determine the response to treatment.
* Patients have blood tests at 3, 6, and 12 months and then annually for 5 years.

DETAILED DESCRIPTION:
Background:

* We have engineered human tumor infiltrating lymphocytes (TIL) and peripheral blood lymphocytes (PBLs) to express a T-cell receptor that recognizes an HLAA 0201 restricted epitope derived from the gp100 protein.
* We constructed a single retroviral vector that contains both Alpha and Beta chains and can mediate genetic transfer of this TCR with high efficiency (greater than 30 percent) without the need to perform any selection.
* In co-cultures with HLA-A*0201 positive melanoma gp100:154-162 TCR transduced T cells secreted significant amount of IFN-Beta (but no significant secretion was observed in control co-cultures with cell lines.
* gp100:154-162 TCR transduced T-cells could efficiently kill HLA-A*0201 positive tumors. There was little or no recognition of normal fibroblasts cells.
* This TCR is over 10 times more reactive with melanoma cells than the MART-1 TCR that mediated tumor regression in two patients with metastatic melanoma.

Objectives:

Primary objectives:

-Determine if the administration of anti-gp100:154-162 TCR-engineered peripheral blood lymphocytes (PBL) or tumor infiltrating lymphocytes (TIL) and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic melanoma.

Secondary objectives:

* Determine the in vivo survival of TCR gene-engineered cells.
* Determine the toxicity profile of this treatment regimen.
* Determine whether treated patients develop anti-mouse TCR antibody.

Eligibility:

Patients who are HLA-A*0201 positive and 18 years of age or older must have

* metastatic melanoma;
* previously received and have been a non-responder to or recurred after aldesleukin
* normal values for basic laboratory values.

Patients may not have:

* concurrent major medical illnesses;
* any form of primary or secondary immunodeficiency;
* severe hypersensitivity to any of the agents used in this study;
* contraindications for high dose aldesleukin administration.

Design:

* If TIL can be obtained and grown but are non-reactive, patients will be assigned to receive TIL transduced with the anti-gp100:154-162 TCR retroviral vector. If TIL cannot be obtained, peripheral blood mononuclear cells (PBMC) will be obtained by leukapheresis (approximately 5 times 10(9) cells) and cultured in the presence of anti-CD3 (OKT3) and aldesleukin and transduced with the antigp100:154-162 TCR retroviral vector. If TIL cells are reactive to autologous tumor or major histocompatibility complex (MHC)-matched tumor cells or PBL cannot be grown, patients will not be treated on this protocol.
* Transduction is initiated by exposure of approximately 10(8) to 5 times 10(8) cells to supernatant containing the anti-gp100:154-162 TCR retroviral vector. These transduced cells will be expanded and tested for their anti-tumor activity.
* Once engineered lymphocytes are demonstrated to be biologically active according to the strict criteria outlined in the Certificate of Analysis, patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, TCR gene-transduced PBMC plus IV aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses).
* Patients will undergo complete evaluation of tumor with physical examination, CT (computed tomography) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met.
* The study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled into each of two cohorts. If 0 or 1 of the 21 patients per cohort experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled in that cohort have a clinical response, then accrual to that cohort will continue until a total of 41 evaluable patients have been enrolled in that cohort.
* The objective will be to determine in two cohorts if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, and anti-gp100:154-162 TCR-gene engineered lymphocytes (TIL and PBL) is able to be associated with a clinical response rate that can rule out 5 percent (p0=0.05) in favor of a modest 20 percent PR (partial response) plus CR (complete response) rate (p1=0.20).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Metastatic melanoma with measurable disease.
  2. Previously received high dose aldesleukin (IL-2) and have been either non-responders (progressive disease) or have recurred.
  3. Positive for gp100 by immunohistochemistry (IHC).
  4. Greater than or equal to 18 years of age.
  5. Willing to sign a durable power of attorney.
  6. Able to understand and sign the Informed Consent Document.
  7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.

     h Life expectancy of greater than three months.

  i. Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.

  j. Must be human leukocyte antigen (HLA-A 0201) positive

  k. Serology:
  1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
  2. Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.

  l. Hematology:
  1. Absolute neutrophil count greater than 1000/mm^3.
  2. White blood cell (WBC) (greater than 3000/ mm^3).
  3. Platelet count greater than 100,000/ mm^3.
  4. Hemoglobin greater than 8.0 g/dl.

  m. Chemistry:
  1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 2.5 times the upper limit of normal.
  2. Serum creatinine less than or equal to 1.6 mg/dl.
  3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

  n. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.

  o. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

  p. Six weeks must have elapsed since prior cytotoxic T-lymphocyte antigen 4 (anti-CTLA4) antibody therapy to allow antibody levels to decline, and patients who have previously received must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Patients with reactive TIL (interferon (IFN)- gamma release greater than 200 pg/mL) available based on overnight co-culture assay with autologous tumor or MHC-matched tumor cells.
2. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
3. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
6. Systemic steroid therapy.
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. History of coronary revascularization.
9. Documented left ventricular ejection faction (LVEF) of less than 45 percent in patients with:

a. Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, 2 degree or 3 degree heart block.

b. Age greater than or equal to 60 years old.

j. Documented forced expiratory volume 1 (FEV1) greater than or equal to 60 percent predicted for patients with:

1. A prolonged history of cigarette smoking (greater than 20 pack/year within the past 2 years).
2. Symptoms of respiratory distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-06; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- [Background] Kawakami Y, Eliyahu S, Sakaguchi K, Robbins PF, Rivoltini L, Yannelli JR, Appella E, Rosenberg SA. Identification of the immunodominant peptides of the MART-1 human melanoma antigen recognized by the majority of HLA-A2-restricted tumor infiltrating lymphocytes. J Exp Med. 1994 Jul 1;180(1):347-52. doi: 10.1084/jem.180.1.347. PMID 7516411
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Sakaguchi K, Appella E, Yannelli JR, Adema GJ, Miki T, Rosenberg SA. Identification of a human melanoma antigen recognized by tumor-infiltrating lymphocytes associated with in vivo tumor rejection. Proc Natl Acad Sci U S A. 1994 Jul 5;91(14):6458-62. doi: 10.1073/pnas.91.14.6458. PMID 8022805
- [Derived] Yao X, Ahmadzadeh M, Lu YC, Liewehr DJ, Dudley ME, Liu F, Schrump DS, Steinberg SM, Rosenberg SA, Robbins PF. Levels of peripheral CD4(+)FoxP3(+) regulatory T cells are negatively associated with clinical response to adoptive immunotherapy of human cancer. Blood. 2012 Jun 14;119(24):5688-96. doi: 10.1182/blood-2011-10-386482. Epub 2012 May 3. PMID 22555974
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0174.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-gp100:154-162 TCR PBL + HD IL-2 | Anti-gp100:154-162 TCR TIL + HD IL-2
Started | 19 | 2
Completed | 19 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-gp100:154-162 TCR PBL + HD IL-2 | Anti-gp100:154-162 TCR TIL + HD IL-2 | Total
Number analyzed (Participants) | 19 | 2 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 2 | 21
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.1 (10.5) | 28.0 (2.8) | 44.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 12 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 2 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 2 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 2 | 21

OUTCOME MEASURES:

1. Primary Outcome: Clinical Tumor Regression.
Description: Clinical tumor regression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is a disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD)is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: 20 months
Measure: Number; unit: Participants
Arm/Group | Anti-gp100:154-162 TCR PBL + HD IL-2 | Anti-gp100:154-162 TCR TIL + HD IL-2
Number analyzed (Participants) | 19 | 2
Participants
  Complete Response | 1 | 0
  Partial Response | 2 | 1
  Progressive Disease | 16 | 1
  Stable Disease | 0 | 0

2. Secondary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 6 years
Measure: Number; unit: Participants
Arm/Group | Anti-gp100:154-162 TCR PBL + HD IL-2 | Anti-gp100:154-162 TCR TIL + HD IL-2
Number analyzed (Participants) | 19 | 2
Participants | 19 | 2

ADVERSE EVENTS:
Arm/Group | Anti-gp100:154-162 TCR PBL + HD IL-2 | Anti-gp100:154-162 TCR TIL + HD IL-2
Serious Adverse Events (participants affected / at risk) | 5/19 | 0/2
Other Adverse Events (participants affected / at risk) | 19/19 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-gp100:154-162 TCR PBL + HD IL-2 (N=19) | Anti-gp100:154-162 TCR TIL + HD IL-2 (N=2)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-gp100:154-162 TCR PBL + HD IL-2 (N=19) | Anti-gp100:154-162 TCR TIL + HD IL-2 (N=2)
Hearing: patients with/without baseline audiogram (Ear and labyrinth disorders) | 8 (8) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 15 (22) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 19 (21) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 19 (22) | 2 (3)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 19 (22) | 2 (3)
Platelets (Blood and lymphatic system disorders) | 18 (18) | 2 (2)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 3 (3) | 0 (0)
Vasovagal episode (Cardiac disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 5 (5) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Constitutional Symptoms-Other (Specify, inability to tolerate IL-2) (General disorders) | 4 (4) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (6) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 2 (2) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16 (17) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhage, GU (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage/Bleeding - Other (hemorrhage) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) (Infections and infestations) | 3 (4) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 3 (3) | 0 (0)
Infection with unknown ANC (Infections and infestations) | 2 (3) | 0 (0)
Febrile neutropenia (Infections and infestations) | 10 (10) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 13 (14) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 8 (10) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Lipase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 7 (9) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arachnoiditis/meningismus/radiculitis (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 6 (6) | 0 (0)
Dizziness (Nervous system disorders) | 8 (8) | 0 (0)
Mood alteration (Nervous system disorders) | 1 (1) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0)
Nystagmus (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 6 (7) | 1 (1)
Vision-blurred vision (Eye disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 3 (6) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute vascular leak syndrome (Vascular disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No